CLINICAL TRIAL: NCT05663762
Title: How do Perceptions of Coronavirus Disease (COVID-19) Risk Influence Health Decisions in Pregnancy?
Status: Completed | Type: Observational
Sponsor: McMaster University (Other)
Collaborators: University of British Columbia (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Other Study IDs: CovPreg2022
Record Dates: First submitted 2022-12-21; First posted 2022-12-23 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Pregnancy Related
Keywords: pregnancy; healthcare use; COVID-19; administrative data; qualitative research
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Pre-pandemic pregnancy and birth: Live hospital births that occurred Jan 1 - Mar 31 2019
- Pregnant and gave birth during the pandemic but before widespread COVID-19 vaccine availability: Live hospital births that occurred Jan 1 - Mar 31 2021
- Pregnant and gave birth during the pandemic and after widespread COVID-19 vaccine availability: Live hospital births that occurred Jan 1 - Mar 31 2022

SUMMARY:
Pregnant people have a higher risk of severe COVID-19 disease. Pregnant people have been disproportionately impacted by COVID-19 infection control policies, which have resulted in higher rates of intimate partner violence, mental health distress, employment and income loss. This project examines the impact of accumulated individual health decisions, describing how perinatal healthcare use and outcomes changed during the COVID-19 pandemic.

Objectives, questions and hypotheses

This research study has two objectives:

1. Describe differences between three groups of pregnant persons classified by the date they gave birth: 01/01/2019-03/31/2019 (2019 birth group), 01/01/2021-03/31/2021 (2021 birth group), and 01/01/2022-03/31/2022 (2022 birth group) pregnancy cohorts in Ontario and British Columbia relative to key outcomes and quality of care indicators related to vaccination, perinatal care, and mental health. Examine the differential impacts on racialized and low-income pregnant people. (Quantitative strand)
2. Understand how pregnant people's perceptions of COVID-19 risk and pandemic circumstances influenced their decision-making about key elements of pregnancy, including vaccination, perinatal care, social support and mental health. (Qualitative strand)

Research questions and hypotheses have been operationalized according to our three themes:

Theme 1: Vaccination Theme 2: Perinatal Care Theme 3: Mental Health and Social Support

DETAILED DESCRIPTION:
This project examines individual health decisions that occur within these structural environments, describing their accumulated impact on key pregnancy outcomes and care indicators related to three themes: vaccination, perinatal care, social supports and mental health. The decisions made during pregnancy have longitudinal impacts on the life of the pregnant person, future child, and family.(1) Given evidence of the particularly difficult situations faced by pregnant people, and the importance of these health decisions, it is important to understand how pandemic circumstances have shaped health decision-making. Understanding how and why pregnant people are making health decisions allows for better clinical and social support as the pandemic endures, and will inform future policy planning. This project is a cross-provincial, parallel mixed-methods study, with thematic data integration at the design and interpretation stages. Ontario and British Columbia were chosen as the two provinces of study because they both experienced a significant impact from COVID-19, both have access to comprehensive administrative health data, and a large number of live births each year.

This study was funded in late February 2022. The quantitative cohort creation plans and data access requests were finalized in late Fall 2022. Qualitative data collection was piloted in Summer 2022, data collection was complete in both provinces August 2023. Study completion is anticipated for February 2024.

ELIGIBILITY:
Inclusion Criteria:

* live, in-hospital birth during the investigators' timeframes of interest
* valid birth date or death date in administrative records
* be of female sex
* been eligible for Ontario Health Insurance Plan in Ontario or Medical Services Plan in British Columbia for the entirety of their pregnancy period

Exclusion Criteria:

* birth outside of a hospital
* stillbirth

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Our total population of Jan 1-Mar 31 births over the three-year study period is therefore approximately 105,000 in Ontario and 31,500 in British Columbia.
Sampling Method: Non-Probability Sample
Enrollment: 136500 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Vaccination | Specified groups from Jan 1 2019 to March 31 2022 (Tdap); Specified groups from Jan 1 2022 to March 31 2022 (Covid-19)
  Were rates of Tdap vaccination different between 2019, 2021, and 2022 birth groups? Outcomes: Tdap (Ontario only) and COVID-19 vaccination rates
Perinatal Care | Specified groups from Jan 1 2019 to March 31 2022
  Were rates of in-person perinatal care different between 2019, 2021, and 2022 birth groups? Outcomes: Gestational diabetes screening, post-partum length of stay
Mental Health and Social Support | Specified groups from Jan 1 2019 to March 31 2022
  Were the rates of clinical diagnosis for new depression, anxiety, and adjustment disorders during pregnancy different between 2019, 2021, and 2022 birth groups?

CONTACTS AND LOCATIONS:
Overall Officials: Meredith Vanstone, PhD, Principal Investigator — McMaster University
Locations (2):
- Canada (2):
  - University of British Columbia, Vancouver, British Columbia
  - McMaster University, Hamilton, Ontario

REFERENCES:
- [Background] Rockliffe L, Peters S, Heazell AEP, Smith DM. Factors influencing health behaviour change during pregnancy: a systematic review and meta-synthesis. Health Psychol Rev. 2021 Dec;15(4):613-632. doi: 10.1080/17437199.2021.1938632. Epub 2021 Jun 29. PMID 34092185
- [Background] Vanstone M, Correia RH, Howard M, Darling E, Bayrampour H, Carruthers A, Davis A, Hadid D, Hetherington E, Jones A, Kandasamy S, Kuyvenhoven C, Liauw J, McDonald SD, Mniszak C, Molinaro ML, Pahwa M, Patel T, Sadik M, Sanya N, Shen K, Greyson D. How do perceptions of Covid-19 risk impact pregnancy-related health decisions? A convergent parallel mixed-methods study protocol. PLoS One. 2023 Aug 10;18(8):e0288952. doi: 10.1371/journal.pone.0288952. eCollection 2023. PMID 37561748
- [Derived] Correia RH, Greyson D, Kirkwood D, Darling EK, Pahwa M, Bayrampour H, Jones A, Kuyvenhoven C, Liauw J, Vanstone M. New perinatal mental health conditions diagnosed during COVID-19: a population-based, retrospective cohort study of birthing people in Ontario. Arch Womens Ment Health. 2025 Aug;28(4):881-894. doi: 10.1007/s00737-024-01534-1. Epub 2024 Nov 19. PMID 39560777
- [Derived] Greyson D, Correia R, Howard M, Darling EK, Kirkwood D, Davis A, Mniszak C, Jones A, Molinaro M, Vanstone M. SARS-CoV-2, Tdap, and influenza vaccination during pregnancy from 2019 to 2022 in Ontario, Canada: a population-based retrospective cohort study. CMAJ. 2024 Sep 30;196(32):E1100-E1113. doi: 10.1503/cmaj.231522. PMID 39353631